CLINICAL TRIAL: NCT04131556
Title: A Phase 1, Open-label, Randomized, Crossover, Bioavailability, Dose Proportionality, and Food Effect Study Comparing the Pharmacokinetics and Palatability of Two Candidate Pediatric Powder-for-Oral-Suspension Formulations of Maribavir to the Current Maribavir Tablet Formulation Administered in Healthy Adult Subjects
Brief Title: A Study Comparing the Pharmacokinetics and Palatability of Two Candidate Pediatric Powder-for-Oral-Suspension Formulations of Maribavir to the Current Maribavir Tablet Formulation Administered in Healthy Adult Participants
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was stopped because based on the planned interim analysis of the data of Part 1, palatability of both pediatric formulations was not acceptable.
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: TAK-620-1019
Record Dates: First submitted 2019-10-17; First posted 2019-10-18 (Actual); Results first posted 2021-01-19 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — maribavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Part 1: Sequence ABC (Experimental): Participants will receive 200 milligram (mg) of maribavir tablet orally (Sequence A) on Day 1 followed by 200 mg maribavir powder for oral suspension with 32.5 percent (%) drug loading (Sequence B) on Day 4 followed by maribavir 200 mg powder for oral suspension with 36.1% drug loading (Sequence C) on Day 7 with a washout period of minimum 72 hours and maximum of 73 hours between Day 1, 4 and 7.
  Interventions: Drug: Maribavir
- Part 1: Sequence BCA (Experimental): Participants will receive 200 mg maribavir powder for oral suspension with 32.5 % drug loading (Sequence B) on Day 1 followed by maribavir 200 mg powder for oral suspension with 36.1% drug loading (Sequence C) on Day 4 and followed by 200 mg of maribavir tablet orally (Sequence A) on Day 7 with a washout period of minimum 72 hours and maximum of 73 hours between Day 1, 4 and 7.
  Interventions: Drug: Maribavir
- Part 1: Sequence CAB (Experimental): Participants will receive maribavir 200 mg powder for oral suspension with 36.1% drug loading (Sequence C) on Day 1 followed by 200 mg of maribavir tablet orally (Sequence A) on Day 4 and followed by 200 mg maribavir powder for oral suspension with 32.5 % drug loading (Sequence B) on Day 7 with a washout period of minimum 72 hours and maximum of 73 hours between Day 1, 4 and 7.
  Interventions: Drug: Maribavir
- Part 1: Sequence CBA (Experimental): Participants will receive maribavir 200 mg powder for oral suspension with 36.1% drug loading (Sequence C) on Day 1 followed by 200 mg maribavir powder for oral suspension with 32.5 percent (%) drug loading (Sequence B) on Day 4 and followed by 200 mg of maribavir tablet orally (Sequence A) on Day 7 with a washout period of minimum 72 hours and maximum of 73 hours between Day 1, 4 and 7.
  Interventions: Drug: Maribavir
- Part 1: Sequence ACB (Experimental): Participants will receive 200 mg of maribavir tablet orally (Sequence A) on Day 1 followed by maribavir 200 mg powder for oral suspension with 36.1% drug loading (Sequence C) on Day 4 and followed by 200 mg maribavir powder for oral suspension with 32.5 % drug loading (Sequence B) on Day 7 with a washout period of minimum 72 hours and maximum of 73 hours between Day 1, 4 and 7.
  Interventions: Drug: Maribavir
- Part 1: Sequence BAC (Experimental): Participants will receive 200 mg maribavir powder for oral suspension with 32.5 % drug loading (Sequence B) on Day 1 followed by 200 mg of maribavir tablet orally (Sequence A) on Day 4 and followed by maribavir 200 mg powder for oral suspension with 36.1% drug loading (Sequence C) on Day 7 and with a washout period of minimum 72 hours and maximum of 73 hours between Day 1, 4 and 7.
  Interventions: Drug: Maribavir
- Part 2: Sequence DEGF (Experimental): Participants under fast will receive 50 mg of maribavir powder for oral suspension (Sequence D) on Day 1 followed by 100 mg of maribavir powder for oral suspension (Sequence E) on Day 4 followed by participants feed with a high fat meal will receive 200 mg of maribavir powder for oral suspension (Sequence G) on Day 7 and then followed by participants under fast will receive 200 mg of maribavir powder for oral suspension (Sequence F) on Day 10 with a washout period of minimum 72 hours and maximum of 73 hours between Day 1, 4, 7 and 10. Doses to be evaluated in Part 2 may be adjusted based on relative bioavailability of the selected pediatric formulation (powder for oral suspension) to the Phase 3 tablet formulation observed in Part 1.
  Interventions: Drug: Maribavir
- Part 2: Sequence EFDG (Experimental): Participants under fast will receive 100 mg of maribavir powder for oral suspension (Sequence E) on Day 1 followed by 200 mg of maribavir powder for oral suspension (Sequence F) on Day 4 followed by 50 mg of maribavir powder for oral suspension (Sequence D) on Day 7 and then followed by participants feed with a high fat meal will receive 200 mg of maribavir powder for oral suspension (Sequence G) on Day 10 with a washout period of minimum 72 hours and maximum of 73 hours between Day 1, 4, 7 and 10. Doses to be evaluated in Part 2 may be adjusted based on relative bioavailability of the selected pediatric formulation (powder for oral suspension) to the Phase 3 tablet formulation observed in Part 1.
  Interventions: Drug: Maribavir
- Part 2: Sequence FGED (Experimental): Participants under fast will receive 200 mg of maribavir powder for oral suspension (Sequence F) on Day 1 followed by participants feed with a high fat meal will receive 200 mg of maribavir powder for oral suspension (Sequence G) on Day 4 followed by participants under fast will receive 100 mg of maribavir powder for oral suspension (Sequence E) on Day 7 and then followed by 50 mg of maribavir powder for oral suspension (Sequence D) on Day 10 with a washout period of minimum 72 hours and maximum of 73 hours between Day 1, 4, 7 and 10. Doses to be evaluated in Part 2 may be adjusted based on relative bioavailability of the selected pediatric formulation (powder for oral suspension) to the Phase 3 tablet formulation observed in Part 1.
  Interventions: Drug: Maribavir
- Part 2: Sequence GDFE (Experimental): Participants feed with a high fat meal will receive 200 mg of maribavir powder for oral suspension (Sequence G) on Day 1 followed by participants under fast will receive 50 mg of maribavir powder for oral suspension (Sequence D) on Day 4 followed by 200 mg of maribavir powder for oral suspension (Sequence F) on Day 7 and then followed by 100 mg of maribavir powder for oral suspension (Sequence E) on Day 10 with a washout period of minimum 72 hours and maximum of 73 hours between Day 1, 4, 7 and 10. Doses to be evaluated in Part 2 may be adjusted based on relative bioavailability of the selected pediatric formulation (powder for oral suspension) to the Phase 3 tablet formulation observed in Part 1.
  Interventions: Drug: Maribavir

INTERVENTIONS:
Drug: Maribavir — Participants in both part 1 and part 2 of the study will receive maribavir tablet or suspension orally depending upon the treatment sequence allocation for a total of 7 and 10 days respectively.
  Other Names: TAK620; SHP620

SUMMARY:
The Purpose of this study is to assess the relative bioavailability, dose proportionality, the impact of food on the rate and extent of absorption, palatability of the selected pediatric formulation of maribavir and the safety and tolerability of two candidate pediatric formulations and the adult tablet formulation of maribavir in healthy participants.

DETAILED DESCRIPTION:
The study will be conducted in two parts (Part 1 and Part 2). Part 1 consists of three treatment periods in six sequences and part 2 consists of four treatment periods in four sequences. In Part 1 two pediatric candidate powder formulations will be compared with maribavir 200mg tablet under fasted conditions in regards to their bioavailability and palatability. In Part 2 dose proportionality and impact of food (a high-fat meal) on the rate and extent of absorption of the selected pediatric formulation will be assessed. The pediatric formulation which will be evaluated in Part 2 will be chosen based on the results of planned analysis of Part 1 PK and palatability data from two candidate pediatric formulations and the doses to be evaluated in Part 2 may be adjusted based on relative bioavailability of the selected pediatric formulation (powder for oral suspension) to the Phase 3 tablet formulation observed in Part 1.

ELIGIBILITY:
Inclusion Criteria:

* An understanding, ability, and willingness to fully comply with study procedures and restrictions.
* Ability to voluntarily provide written, signed, and dated (personally or via a legally-authorized representative) informed consent/and assent as applicable to participate in the study.
* Age 18-50 years, inclusive at the time of consent.
* Male, or non-pregnant, non-breastfeeding female who agrees to comply with any applicable contraceptive requirements of the protocol or females of non-childbearing potential.
* Healthy as determined by the investigator on the basis of screening evaluations.
* Hemoglobin for males greater than or equal to (> or =)135.0 gram per liter (g/L) and females > or = 120.0 g/L at screening and on Day -1.
* Body mass index (BMI) between 18.0 and 30.0 kilogram per meter square (kg/m2) inclusive with a body weight greater than (>) 50 kg (110 lbs).

Exclusion Criteria:

* History of any hematological, hepatic, respiratory, cardiovascular, renal, neurological or psychiatric disease, gallbladder removal, or current recurrent disease.
* Current or relevant history of physical or psychiatric illness, any medical disorder that may require treatment or make the participant unlikely to fully complete the study, or any condition that presents undue risk from the investigational product or procedures.
* Known or suspected intolerance or hypersensitivity to the investigational product(s), closely-related compounds, or any of the stated ingredients.
* Significant illness, as judged by the investigator, within 2 weeks of the first dose of investigational product.
* Donation of blood or blood products (e.g., plasma or platelets) within 60 days prior to receiving the first dose of investigational product.
* Within 30 days prior to the first dose of investigational product:a) Have used an investigational product, b) Have been enrolled in a clinical study (including vaccine studies) that, in the investigator's opinion, may impact this study, c) Have had any substantial changes in eating habits, as assessed by the investigator.
* Confirmed systolic blood pressure >139 millimetre of mercury (mmHg) or < 89 mmHg, and diastolic blood pressure > 89 mmHg or < 49 mmHg.
* Twelve-lead ECG demonstrating QTc > 450 millisecond (msec).
* Known history of alcohol or other substance abuse within the last year.
* Male participants who consume more than 21 units of alcohol per week or 3 units per day. Female participants who consume more than 14 units of alcohol per week or 2 units per day.
* A positive screen for alcohol or drugs of abuse at screening or on Day -1 of Treatment Period.
* A positive human immunodeficiency virus (HIV), HBsAg, or Hepatitis C virus (HCV) antibody screen.
* Use of tobacco in any form (e.g., smoking or chewing) or other nicotine-containing products in any form (e.g., gum, patch).
* Routine consumption of more than 2 units of caffeine per day or participants who experience caffeine withdrawal headaches.
* Prior screen failure, randomization, enrollment, participation in this study or participation in Part 1 of this study.
* Current use of any prescription medication with the exception of hormonal replacement therapy. (Current use is defined as use within 30 days of the first dose of investigational product.) Current use of any over the counter medication (including herbal, or homeopathic preparations) within 14 days of the first dose of investigational product.
* Current use of antacids and H2 antagonists.
* Ingestion of known CYP3A modulators within 7 days of Day 1, Period 1.
* Inability or unwillingness to consume 100 percent of high-fat meal in Part 2 (including participants with lactose or gluten intolerance).
* History of oral/nasal cavity infections, gastroesophageal reflux, asthma treatment with albuterol, zinc supplementation.
* Participants with dry mouth syndrome or burning mouth syndrome or menopausal women suffering from dysgeusia.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-10-25 (Actual); Primary Completion 2020-01-06 (Actual); Study Completion 2020-01-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Shire
Locations (1):
- Clinical Pharmacology of Miami, Llc, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data from this particular study will not be shared as the data are subject to contractual (or consent) provisions that prohibit transfer to third parties.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at single site in United States of America from 25 October 2019 (first participant first visit) and 06 January 2020 (last participant last visit).
Pre-assignment Details: This study was planned to be conducted in 2 parts: Part 1 and Part 2. However, study was terminated based on planned interim analysis of the data of Part 1, palatability of both pediatric formulations was not acceptable and therefore, Part 2 was not conducted. Participants were randomized to 1 of 6 sequences with treatment A, B and C. Baseline characteristics of participants were only analyzed and reported for overall study period, as planned, and not per treatment to avoid double-counting.
Groups:
- Maribavir: Participants received 200 milligrams (mg) of maribavir tablet orally (Treatment A) or 200 mg maribavir powder for oral suspension with 32.5 percent (%) drug loading (Treatment B) or maribavir 200 mg powder for oral suspension with 36.1% drug loading (Treatment C) on Day 1 or Day 4 or Day 7 in different sequences of ABC, BCA, CAB, CBA, ACB, and BAC.
Period: Overall Study
Arm/Group | Maribavir
Started | 20
Completed | 18
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Safety set 1 consisted of all participants who received at least 1 dose of maribavir in Part 1.
Arm/Group | Maribavir
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: Years] | 33.7 (8.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Maximum Concentration (Cmax) Occurred at Time of Maximum Observed Concentration Sampled During a Dosing Interval (Tmax) of Maribavir in Plasma
Description: Cmax defined as maximum concentration occurred at tmax of maribavir in plasma was reported. Geometric mean and geometric coefficient of variation percent (CV%) were reported.
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16, 20, 24 hours post-dose on Days 1, 4, and 7
Population: Pharmacokinetic (PK) set 1 consisted of participants who received at least 1 dose of maribavir, did not vomit within 4 hours post dosing, and had at least 1 evaluable post-dose maribavir concentration value in Part 1. Data for the PK parameters were planned and analyzed based on unique treatment sequence A, B, C. Hence, data was reported separately.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micrograms per milliliter (mcg/mL)
Groups:
- Treatment A: Participants received 200 milligrams (mg) of maribavir tablet orally on Day 1 or Day 4 or Day 7.
- Treatment B: Participants received 200 mg maribavir powder for oral suspension with 32.5 percent (%) drug loading on Day 1 or Day 4 or Day 7.
- Treatment C: Participants received maribavir 200 mg powder for oral suspension with 36.1% drug loading on Day 1 or Day 4 or Day 7.
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 18 | 19 | 20
Micrograms per milliliter (mcg/mL) | 10.7 (31.42) | 7.35 (46.92) | 6.84 (56.71)
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; Test type: Equivalence — Equivalence analysis based on confidence intervals (CIs). If the 90% CIs of the geometric mean ratios were within (0.8, 1.25), bioequivalence between the two formulations (test powder for oral suspension versus reference tablet) was to be claimed. A linear mixed effect ANOVA model with treatment, period, sequence as fixed effects and participant within sequence as a random effect was used to fit to ln-transformed PK parameters; ANOVA; % Ratio of Geometric least square means = 67.76, 90% CI 2-sided [59.50 to 77.16]
Statistical Analysis 2: Comparison: Treatment A vs Treatment C; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; % Ratio of Geometric least squares means = 62.29, 90% CI 2-sided [54.73 to 70.90]

2. Primary Outcome: Part 1: Time of Maximum Observed Concentration Sampled During a Dosing Interval (Tmax) of Maribavir in Plasma
Description: tmax defined as time of maximum observed concentration sampled during a dosing interval of maribavir in plasma were reported.
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16, 20, 24 hours post-dose on Days 1, 4, and 7
Population: PK set 1 consisted of participants who received at least 1 dose of maribavir, did not vomit within 4 hours post dosing, and had at least 1 evaluable post-dose maribavir concentration value in Part 1. Data for the PK parameters were planned and analyzed based on unique treatment sequence A, B, C. Hence, data was reported separately.
Measure: Median (Full Range); unit: Hour
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 18 | 19 | 20
Hour | 1.00 [0.500 to 2.00] | 3.00 [1.00 to 4.00] | 2.00 [1.00 to 4.00]
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; Statistical analysis of tmax was performed using a nonparametric test. The median difference of tmax between treatments and 90% CIs of the median differences were calculated from Hodges-Lehman estimate, and p-value was produced from Wilcoxon signed rank test; Test type: Other; p < .001, Wilcoxon signed rank test; Median Difference (Final Values) = 1.25, 90% CI 2-sided [0.75 to 1.75]
Statistical Analysis 2: Comparison: Treatment A vs Treatment C; [analysis description as in outcome 2, analysis 1]; Test type: Other; p < .001, Wilcoxon signed rank test; Median Difference (Final Values) = 1.00, 90% CI 2-sided [0.75 to 1.25]

3. Primary Outcome: Part 1: Area Under the Curve From the Time of Dosing to the Last Measurable Concentration (AUC0-last) of Maribavir in Plasma
Description: AUC0-last of maribavir in plasma was reported. Geometric mean and geometric coefficient of variation percent (CV%) were reported.
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16, 20, 24 hours post-dose on Days 1, 4, and 7
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*micrograms per milliliter (h*μg/mL)
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 18 | 19 | 20
Hour*micrograms per milliliter (h*μg/mL) | 50.1 (49.21) | 41.2 (55.09) | 39.1 (60.58)
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; % Ratio of Geometric least squares means = 81.27, 90% CI 2-sided [73.88 to 89.40]
Statistical Analysis 2: Comparison: Treatment A vs Treatment C; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; % Ratio of Geometric least squares means = 78.00, 90% CI 2-sided [70.92 to 85.79]

4. Primary Outcome: Area Under the Curve Extrapolated to Infinity, Calculated Using the Observed Value of the Last Non-Zero Concentration (AUC0-Inf) of Maribavir in Plasma
Description: AUC0-Inf of maribavir in plasma was reported. Geometric mean and geometric coefficient of variation percent (CV%) were reported.
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16, 20, 24 hours post-dose on Days 1, 4, and 7
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*μg/mL
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 18 | 19 | 20
h*μg/mL | 52.5 (49.72) | 44.5 (56.26) | 42.4 (60.69)
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; % Ratio of Geometric least squares means = 83.52, 90% CI 2-sided [76.12 to 91.64]
Statistical Analysis 2: Comparison: Treatment A vs Treatment C; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; ANOVA; % Ratio of Geometric least squares means = 80.36, 90% CI 2-sided [73.26 to 88.16]

5. Primary Outcome: Part 1: Terminal Half-Life (t1/2) of Maribavir in Plasma
Description: t1/2 of maribavir in plasma was reported.
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16, 20, 24 hours post-dose on Days 1, 4 and 7
Population: as for outcome 2
Measure: Median (Full Range); unit: Hour
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 18 | 19 | 20
Hour | 4.04 [1.33 to 8.07] | 4.80 [1.90 to 11.6] | 5.95 [1.36 to 10.1]

6. Primary Outcome: Part 1: Apparent Total Body Clearance Following Extravascular Administration (CL/F) of Maribavir in Plasma
Description: CL/F of maribavir in Plasma was reported.
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16, 20, 24 hours post-dose on Days 1, 4 and 7
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Liters per hour (L/h)
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 18 | 19 | 20
Liters per hour (L/h) | 4.21 (1.99) | 5.13 (2.82) | 5.49 (3.29)

7. Primary Outcome: Part 1: Delay Between the Time of Dosing and Time of Appearance of Plasma Concentration (Tlag) of Maribavir in Plasma
Description: Tlag of maribavir in plasma was reported.
Time Frame: Pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 12, 16, 20, 24 hours post-dose on Day 1, 4 and 7
Population: as for outcome 2
Measure: Median (Full Range); unit: Hour
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 18 | 19 | 20
Hour | 0.00 [0.00 to 0.250] | 0.250 [0.00 to 0.500] | 0.250 [0.00 to 0.500]
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; Statistical analysis of Tlag was performed using a nonparametric test. The median difference of Tlag between treatments and 90% CIs of the median differences were calculated from Hodges-Lehman estimate, and p-value was produced from Wilcoxon signed rank test; Test type: Other; p = 0.006, Wilcoxon signed rank test; Median Difference (Final Values) = 0.13, 90% CI 2-sided [0.13 to 0.25]
Statistical Analysis 2: Comparison: Treatment A vs Treatment C; [analysis description as in outcome 7, analysis 1]; Test type: Other; p = 0.011, Wilcoxon signed rank test; Median Difference (Final Values) = 0.13, 90% CI 2-sided [0.13 to 0.25]

8. Primary Outcome: Part 1: Number of Participants With Responses to Palatability Assessment up to Day 7
Description: The palatability was evaluated to identify, characterize and quantify the sensory attributes of products, e.g., basic tastes, texture and mouth feel and to assess the overall acceptability. Number of participants responded to palatability assessment up to Day 7 were reported.
Time Frame: Up to Day 7
Population: Safety set 1 consisted of all participants who received at least 1 dose of maribavir in Part 1. Data for the palatability was planned and analyzed based on unique treatment sequence A, B, C. Hence, data was reported separately.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 18 | 19 | 20
Participants
  How this drug tasted to you?: Bitter | 2 | 14 | 14
  How this drug tasted to you?: Salty | 0 | 0 | 1
  How this drug tasted to you?: Sour | 0 | 1 | 0
  How this drug tasted to you?: Sweet | 0 | 0 | 0
  How this drug tasted to you?: Savory | 0 | 0 | 0
  How this drug tasted to you?: No taste | 16 | 4 | 5
  How strong was the taste?: Strong | 0 | 8 | 8
  How strong was the taste?: Medium | 1 | 6 | 3
  How strong was the taste?: Weak | 1 | 1 | 4
  How strong was the taste?: no taste | 16 | 4 | 5
  Did the drug have a rough or gritty texture?: No | 18 | 4 | 4
  Did the drug have a rough or gritty texture?: Yes | 0 | 15 | 16
  Was the drug easy to swallow?: No | 0 | 0 | 0
  Was the drug easy to swallow?: Yes | 18 | 19 | 20
  Overall taste & texture?: Agree | 18 | 10 | 13
  Overall taste & texture?: Neither agree/disagree | 0 | 5 | 4
  Overall taste & texture?: Disagree | 0 | 4 | 3

9. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product and that does not necessarily had a causal relationship with this treatment. A TEAE was an adverse event with a start date on or after the first dose of Investigational product (IP), or a start date before the date of the first dose of IP but increased in severity on or after the date of the first dose of IP. Number of participants with TEAEs were reported.
Time Frame: From start of study drug administration up to follow-up (Day 17)
Population: Safety Set 1 consisted of all participants who received at least 1 dose of maribavir in Part 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Maribavir
Number analyzed (Participants) | 20
Participants | 3

10. Secondary Outcome: Number of Participants With Clinically Significant Changes in Vital Signs Reported as TEAEs
Description: Vital sign assessments included systolic and diastolic blood pressure, pulse rate and body temperature. Any change in vital signs which were deemed clinically significant by the investigator were recorded as TEAE.
Time Frame: From start of study drug administration up to follow-up (Day 17)
Population: Safety set 1 consisted of all participants who received at least 1 dose of maribavir in Part 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Maribavir
Number analyzed (Participants) | 20
Participants | 0

11. Secondary Outcome: Number of Participants With Clinically Significant Changes in Electrocardiogram (ECG) Reported as TEAEs
Description: 12-lead ECG were evaluated. Any change in ECG assessments which are deemed clinically significant by the investigator were reported as TEAE.
Time Frame: From start of study drug administration up to follow-up (Day 17)
Population: Safety set 1 consisted of all participants who received at least 1 dose of maribavir in Part 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Maribavir
Number analyzed (Participants) | 18
Participants | 0

12. Secondary Outcome: Number of Participants With Clinically Significant Changes in Clinical Laboratory Results Reported as TEAEs
Description: Clinical laboratory tests included biochemistry, hematology and urinalysis. Any change in clinical laboratory results which are deemed clinically significant by the investigator were reported as TEAE.
Time Frame: From start of study drug administration up to follow-up (Day 17)
Population: Safety set 1 consisted of all participants who received at least 1 dose of maribavir in Part 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Maribavir
Number analyzed (Participants) | 18
Participants | 0

ADVERSE EVENTS:
Time Frame: From start of study drug administration up to follow-up (Day 17)
Arm/Group | Maribavir
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 3/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Maribavir (N=20)
Flatulence (Gastrointestinal disorders) | 1 (1)
Liver function test increased (Investigations) | 1 (1)
Headache (Nervous system disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Sponsor terminated this study based on the planned interim analysis of the data of Part 1, palatability of both pediatric formulations was not acceptable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.

DOCUMENTS (2):
  • Study Protocol (2019-11-05): https://cdn.clinicaltrials.gov/large-docs/56/NCT04131556/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-18): https://cdn.clinicaltrials.gov/large-docs/56/NCT04131556/SAP_001.pdf